CLINICAL TRIAL: NCT03411408
Title: Accelerated Hypofractionated Intensity - Modulated Radiotherapy After Hyperbaric Oxygenation for Recurrent High Grade Glioma: a Pilot Study
Brief Title: Accelerated Hypofractionated Intensity - Modulated Radiotherapy After Hyperbaric Oxygenation for Recurrent High Grade Glioma.
Acronym: HBO-RT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST191.02
Record Dates: First submitted 2018-01-11; First posted 2018-01-26 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Malignant Glioma; High Grade Glioma; Recurrent Glioma
Keywords: Hypofractionated radiotherapy; image - guided helical tomotherapy; hyperbaric oxygen therapy; malignant glioma; high grade glioma; recurrent glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HBO and RT (Experimental): Hyperbaric oxygenation therapy and Accelerated Hypofractionated intensity - modulated radiotherapy
  Interventions: Device: HBO; Radiation: RT

INTERVENTIONS:
Device: HBO — Hyperbaric oxygen is administrated in a multiplace hyperbaric chamber according to the following schedule:
  Ten minutes of compression with a Fraction of inspired oxygen (FiO2) more than 90% from 152 to 253 kilopascal, 60 minutes of Fraction of inspired oxygen (FiO2) more than 90% at 253 kilopascal (three breathing cycles in oxygen for 22 minutes each, with two intervals breathing air for 2 minutes each) and 10 minutes of decompression with a Fraction of inspired oxygen (FiO2) more than 90% from 253 to 152 kilopascal.
Radiation: RT — tomotherapy (within 60 minutes from completion of decompression of hyperbaric chamber) with 3-5 consecutive sessions- one fraction per day, 5 Gy / die .

SUMMARY:
This is a pilot study of radiotherapy using Hypofractionated image - guided helical tomotherapy after hyperbaric oxygen HBO therapy for treatment of recurrent malignant High-grade gliomas. HBO therapy will be perform in conjunction with each RT session.

The treatment scheme is:

Hyperbaric oxygenation therapy (the maximum period of time from completion of decompression to RT is 60 min) followed by tomotherapy (3-5 consecutive sessions- one fraction per day , 5 Gy / die ).

The trial will enroll 24 patients in 24 months with a follow-up period of 1 year.

DETAILED DESCRIPTION:
This is a pilot study to evaluate the efficacy of hypofractionated image- guided helical tomotherapy after hyperbaric oxygen therapy (HBO) for treatment of recurrent malignant high - grade gliomas The primary objective of this study is to evaluate the disease control rate (DCR) of treated patients.

The secondary Objectives are:

* Safety assessment (acute and late toxicity).
* Overall Survival (OS),
* Progression Free Survival (PFS).
* Evaluation of predictive score of disease, radionecrosis and pseudoprogression using perfusion DSC and DCE MRI

Patients will receive fractionated stereotactic radiotherapy using tomotherapy combined with hyperbaric oxygen (HBO) therapy.

Hyperbaric oxygenation therapy (the maximum period of time from completion of decompression to RT is 60 min) followed by tomotherapy (3-5 consecutive sessions- one fraction per day, 5 Gy / die).

The overall duration of treatment will be max 5 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, aged >18 years.
2. Karnofsky Performance Scale (KPS)> 60
3. Imaging confirmation of first tumor progression o regrowth as defined by Response Assessment in Neuro-Oncology Criteria (RANO) criteria at least 12 weeks after completion of radiotherapy, unless the recurrence is outside the radiation field or has been histologically documented
4. Recurrence after adjuvant treatment( surgery followed by radiotherapy and chemotherapy) in patients who could receive further therapeutic interventions
5. No more than one prior line of chemotherapy (one line of chemotherapy after concurrent and adjuvant Temozolomide (TMZ) - based chemotherapy or procarbazine/lomustine/vincristine (PCV) - Radiotherapy (RT)
6. Patients who have undergone recent surgery for recurrent o progressive high grade gliomas are eligible provided that : surgery must have confirmed the recurrence ; a minimum of 28 days must have elapsed from the days of surgery to study . For core or needle biopsy a minimum of 7 days must have elapsed prior to study .
7. If female and of child bearing potential , have a negative result on a pregnancy test performed a maximum of 7 days before initiation .
8. Female participants of child bearing potential and male participants whose partner is of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study and for 4 months thereafter
9. Have adequate bone marrow function , liver function , and renal function , as measured by following laboratory assessments conducted within 7 days prior to the initiation of study treatment .
10. Hemoglobin >9.0 g/dl
11. Absolute neutrophil count (ANC) >1500/mm3 without transfusions or granulocyte colony stimulating factor and other hematopoietic growth factors
12. Platelet count ≥90,000/μl
13. White Blood Cell (WBC) >3.0 x 109/L
14. Total bilirubin <1.5 times the upper limit of normal
15. Serum creatinine <1.5 x upper limit of normal
16. Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

1. Radiotherapy within 12 weeks prior to the diagnosis of progression, if the lesion is in the radiation field.
2. Patients with cardiopulmonary diseases (heart failure, bolus emphysema, pneumothorax, chronic obstructive pulmonary disease (COPD) with hypercapnia sinusitis )
3. Closed angle-glaucoma with pressure ocular superior to 24 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-02-22 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Disease control rate (DCR) | up to one year
  DCR will be evaluated by performing MRI images The treatment response will be evaluated according to the RANO criteria

SECONDARY OUTCOMES:
Incidence of adverse events | up to 36 months
  Adverse events will be graded according to the National Cancer Institute Common Terminology Criteria Events v. 4.03.
Overall survival (OS) | up to 36 months
  OS will be defined as the time from the first day of treatment to death due any cause or censored at date last known alive
Progression Free survival (PFS) | up to 36 months
  PFS will be calculated as the time from the first day of treatment to the date of the first observation of documented disease progression or death due to any cause. Patients without tumor progression at the time of analysis will be censored at their last date of tumor evaluation.
Predictive score of disease progression by DSC MRI | up to 36 months
  determining a predictive score of disease, using perfusion dynamic contrast-enhanced (DSC) permeability MRI
Radionecrosis by DSC MRI | up to 36 months
  determining radionecrosis using perfusion dynamic contrast-enhanced (DSC) permeability MRI
Pseudoprogression by DSC MRI | up to 36 months
  determining pseudoprogression using perfusion dynamic contrast-enhanced (DSC) permeability MRI
Predictive score of disease progression by DCE MRI | up to 36 months
  determining a predictive score of disease using dynamic susceptibility contrast (DCE) perfusion MRI
Radionecrosis by DCE MRI | up to 36 months
  determining radionecrosis using dynamic susceptibility contrast (DCE) perfusion MRI
pseudoprogression by DCE MRI | up to 36 months
  determining pseudoprogression using dynamic susceptibility contrast (DCE) perfusion MRI

CONTACTS AND LOCATIONS:
Overall Officials: Donatella Arpa, Principal Investigator — IRST IRCCS
Locations (3):
- Italy (3):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola, FC
  - Centro Iperbarico, Ravenna, RA
  - Neuroradiology, AUSL della Romagna - RAVENNA, Ravenna, RA

REFERENCES:
- [Derived] Arpa D, Parisi E, Ghigi G, Cortesi A, Longobardi P, Cenni P, Pieri M, Tontini L, Neri E, Micheletti S, Ghetti F, Monti M, Foca F, Tesei A, Arienti C, Sarnelli A, Martinelli G, Romeo A. Role of Hyperbaric Oxygenation Plus Hypofractionated Stereotactic Radiotherapy in Recurrent High-Grade Glioma. Front Oncol. 2021 Mar 30;11:643469. doi: 10.3389/fonc.2021.643469. eCollection 2021. PMID 33859944